CLINICAL TRIAL: NCT04142216
Title: Effect of Chewing Gum on Interdialytic Weight Gain, Thirst, Dry Mouth and Intradialytic Symptoms in Hemodialysis Patients: A Prospective Randomized Controlled Trial
Brief Title: Effect of Chewing Gum in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Nurten Ozen, Assistant Professor, Istanbul Demiroglu Bilim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019/7
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Results first posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Chewing Gum; Hemodialysis
Keywords: Thirst; Weight gain
MeSH Terms: conditions — Weight Gain | interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chewing gum group (Experimental): The patients will be asked to chew on a regular chewing gum for three months.
  Interventions: Dietary Supplement: Chewing Gum
- Control group (No Intervention): The patients will not chewing gum during three months.

INTERVENTIONS:
Dietary Supplement: Chewing Gum — The patients will chew one piece of regular chewing gum six times in a day and feeling of thirst for ten minutes for three months.
  Arms: Chewing gum group

SUMMARY:
The aim of this prospective randomized controlled study was to investigate the effects of chewing gum on interdialytic weight gain, thirst, dry mouth and intradialytic symptoms in hemodialysis patients.

DETAILED DESCRIPTION:
The prevalence of xerostomia varies high in patients with chronic hemodialysis (HD), and the decreased saliva flow rate due to various mechanisms is the main factor in its development. The significant decrease in saliva flow due to the atrophy and fibrosis of the salivary glands in HD patients is further affected by the restriction in fluid intake. The use of drugs such as antidepressants, antipsychotics, antihistamines, antihypertensives, aspirin, benzodiazepines, opioids and proton pump inhibitors also leads to hyposalivation and xerostomia. Thirst is common in chronic HD patients due to both volumetric and osmometric causes but the primary mechanism is osmometric. The osmolarity of the extracellular fluid increases with the dietary salt and the hypothalamus is stimulated by the shrinkage of the osmoreceptor cells, leading to the desire to ingest liquids. Volumetric thirst develops secondary to water and salt loss and the resultant stimulation of cardiac baroreceptors, with the cardiac return volume decreasing gradually towards the end of the HD session. Increased interdialytic weight in HD patients causes increased risk of death due to cerebrovascular events and cardiovascular diseases and leads to an increase in morbidity and mortality together with a deterioration of the patient's quality of life. Interdialytic weight gain (IWG) causes incompliance with fluid control as a result of the secondary excessive consumption of liquid and food and is an important condition.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* On maintenance hemodialysis three times per week for four hours per session
* Receiving hemodialysis therapy for a least six moths at the time of the study
* Able to communicate in Turkish
* Willing to participate to the study

Exclusion Criteria:

* 18 years of age younger
* Absence of psychiatric disorders that cause cognitive dysfunction, such as Alzheimer's disease or chronic psychosis.
* The patient who took chemotherapy and radiotherapy
* Have salivary gland infection and dementia
* Oral and / or dental diseases to prevent chewing gum
* Unwilling to to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Ozen, Asst. Prof, Principal Investigator — Istanbul Demiroglu Bilim University
Locations (1):
- Demiroglu Bilim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bots CP, Brand HS, Veerman EC, Valentijn-Benz M, Van Amerongen BM, Valentijn RM, Vos PF, Bijlsma JA, Bezemer PD, Ter Wee PM, Amerongen AV. Interdialytic weight gain in patients on hemodialysis is associated with dry mouth and thirst. Kidney Int. 2004 Oct;66(4):1662-8. doi: 10.1111/j.1523-1755.2004.00933.x. PMID 15458464
- [Background] Cabrera C, Brunelli SM, Rosenbaum D, Anum E, Ramakrishnan K, Jensen DE, Stalhammar NO, Stefansson BV. A retrospective, longitudinal study estimating the association between interdialytic weight gain and cardiovascular events and death in hemodialysis patients. BMC Nephrol. 2015 Jul 22;16:113. doi: 10.1186/s12882-015-0110-9. PMID 26197758
- [Background] Duruk N, Eser I. The Null Effect of Chewing Gum During Hemodialysis on Dry Mouth. Clin Nurse Spec. 2016 Sep-Oct;30(5):E12-23. doi: 10.1097/NUR.0000000000000234. PMID 27509571
- [Background] Jagodzinska M, Zimmer-Nowicka J, Nowicki M. Three months of regular gum chewing neither alleviates xerostomia nor reduces overhydration in chronic hemodialysis patients. J Ren Nutr. 2011 Sep;21(5):410-7. doi: 10.1053/j.jrn.2010.08.002. Epub 2010 Dec 24. PMID 21185739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: The assignment of patients to groups has began on October 14, 2019. It lasted on November 1, 2019.
Pre-assignment Details: in chewing group: one person reject to join to the study. one person chewing clove.
Period: Overall Study
Arm/Group | Control Group | Chewing Gum Group
Started | 28 | 28
Completed | 22 | 22
Not Completed | 6 | 6
Not completed — Hospitalization | 0 | 2
Not completed — Death | 3 | 1
Not completed — Referral to another hemodialysis unit | 3 | 2
Not completed — Use of clove | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chewing Gum Group | Control Group | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.72 (15.21) | 61.40 (16.64) | 61.56 (15.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 22
  Male | 8 | 14 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Intradialytic Weight Gain
Description: Interdialytic weight gain was defined as the difference between the predialytic weight and weight at the end of the previous dialysis session
Time Frame: up to 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Control Group | Chewing Gum Group
Number analyzed (Participants) | 22 | 22
kg | 2.53 (0.80) | 2.44 (0.95)

2. Primary Outcome: Change From Baseline Feeling of Thirst at Three Months
Description: It will be assessed three times at the end of the dialysis session with Visual Analogue. Thirst intensity measured on a Visual Analog Scale with scores ranging from 0 - 10. Thirst increases as the score increases. The high point describes bad outcome.
Time Frame: At the end of the 1st, 6th, 12th week (3 hemodialysis sessions are done every week)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Chewing Gum Group
Number analyzed (Participants) | 22 | 22
score on a scale | 5.04 (2.76) | 1.72 (2.07)

3. Primary Outcome: Change From Baseline Dry Mouth at Three Months
Description: It will be assessed three times at the end of the dialysis session with Visual Analogue Scale. Visual Analogue Scale ranging from 0 (no dry mouth) to 10 (worst dry mouth). Dry mouth increases the score increases. The high point describes bad outcome.
Time Frame: At the end of the 1st, 6th, 12th week (3 hemodialysis sessions are done every week)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Chewing Gum Group
Number analyzed (Participants) | 22 | 22
units on a scale | 5.04 (2.76) | 1.72 (2.07)

4. Primary Outcome: Change From Baseline Dry Mouth at Three Months
Description: It will be assessed two times at the end of the dialysis session with sample of saliva. Saliva flow rate/minute will be measured. Saliva flow rate/minute is presented with "ml".
Time Frame: At the end of the 1st and 12th week (3 hemodialysis sessions are done every week)
Measure: Mean (Standard Deviation); unit: ml/minute
Arm/Group | Control Group | Chewing Gum Group
Number analyzed (Participants) | 22 | 22
ml/minute | 5.04 (2.76) | 1.72 (2.07)

5. Primary Outcome: Change From Baseline Intradialytic Symptoms at Three Months
Description: It will be assessed with "Dialysis Symptom Index". Using this scoring system, the minimum possible total severity score was 0 if none of the 30 symptoms was present and the maximum potential. Score was 150 if all of the 30 symptoms were reported and rated as "very much bothersome". The minimum value is "0" and the maximum value is "150".
Time Frame: At the end of the 1st and 12th week (3 hemodialysis sessions are done every week)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Chewing Gum Group
Number analyzed (Participants) | 22 | 22
score on a scale | 19.13 (13.71) | 19.18 (15.27)

6. Secondary Outcome: Change From Baseline Anxiety at Three Months
Description: It will be assessed with Hospital Anxiety and Depression Scale. This scale, which has a two-factor structure is comprised of 14 items. Seven of these items assess the anxiety status and the remaining seven assess depression. Each item is scored on a four-point scale. Total score ranges between 0 and 21 for anxiety and depression. Scores between 0 and 7 indicate normal emotional status.
Time Frame: At the end of the 1st and 12th week (3 hemodialysis sessions are done every week)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Chewing Gum Group
Number analyzed (Participants) | 22 | 22
score on a scale | 8.18 (5.50) | 8.40 (5.71)

7. Secondary Outcome: Change From Baseline Fluid Control at Three Months
Description: It will be assessed with "Fluid Control Scale in Hemodialysis Patients". the scale had 24 items and three subdimensions,namely, knowledge, behavior, and attitude. The lowest score obtained from the scale was 24 and the highest score was 72, and the higher the score, the greater the compliance of the patients with fluid control.
Time Frame: At the end of the 1st and 12th week (3 hemodialysis sessions are done every week)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Chewing Gum Group
Number analyzed (Participants) | 22 | 22
score on a scale | 53.95 (6.06) | 58.04 (4.82)

8. Secondary Outcome: Change From Baseline Depression at Three Months
Description: as for outcome 6
Time Frame: At the end of the 1st and 12th week (3 hemodialysis sessions are done every week)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Chewing Gum Group
Number analyzed (Participants) | 22 | 22
score on a scale | 8.63 (4.90) | 8.13 (4.31)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks.
Description: Side effects were not monitored.
Arm/Group | Control Group | Chewing Gum Group
All-Cause Mortality (participants affected / at risk) | 3/28 | 1/28
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT04142216/Prot_SAP_000.pdf